CLINICAL TRIAL: NCT05487196
Title: Effectiveness of Clonidine, Dexmedetomidine, and Fentanyl Adjuncts for Labor Epidural Analgesia: A Randomized Controlled Quadruple Blinded Non-Inferiority Trial (CLASSIER Trial)
Brief Title: Effectiveness of Clonidine, Dexmedetomidine, and Fentanyl Adjuncts for Labor Epidural Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY22030095
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Vaginal Delivery; Epidural Labor Analgesia
MeSH Terms: interventions — Clonidine; Dexmedetomidine; Fentanyl; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, quadruple blinded, parallel arm, controlled, non-inferiority trial in 3 groups allocated in a 1:1:1 ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clonidine (Experimental): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Clonidine 60 mcg
  Interventions: Drug: Clonidine; Drug: Ropivacaine
- Dexmedetomidine (Experimental): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Dexmedetomidine 30 mcg
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine
- Ropivacaine + Fentanyl (Active Comparator): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Fentanyl 100mcg
  Interventions: Drug: Fentanyl; Drug: Ropivacaine

INTERVENTIONS:
Drug: Clonidine — Clonidine belongs to the drug classification of antihypertensives
  Arms: Clonidine
Drug: Dexmedetomidine — Dexmedetomidine belongs to the drug classification of sedatives
  Arms: Dexmedetomidine
Drug: Fentanyl — Fentanyl belongs to the drug classification of analgesic opioid agonists and is used as the standard of care
  Arms: Ropivacaine + Fentanyl
Drug: Ropivacaine — Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care

SUMMARY:
The purpose of this randomized controlled trial is to compare the effectiveness of epidural clonidine, dexmedetomidine, or fentanyl adjuncts for labor analgesia.

DETAILED DESCRIPTION:
Adjuncts for epidural labor analgesia have remained unchanged for decades, whereas changes in patient population and the opioid epidemic have created an increased demand for non-opioid alternative adjuncts to limit peripartum opioid exposure. This study aims to identify effective alternative and non-opioid adjunctive agents for epidural labor analgesia.

The opioid crisis in the United States has translated to an increasing number of pregnant women requiring care for labor and delivery. These trends have resulted in new questions about alternative epidural analgesia adjuncts besides lipophilic opioids (e.g., fentanyl and sufentanil) because: 1) many people with opioid or substance use disorder desire to avoid opioids in all formulations and routes of administration; and 2) epidural fentanyl or sufentanil administration for labor can potentially interfere with the accuracy of urine drug screening in the postpartum period, which has implications for postpartum social services considerations.

Some existing literature suggests that dexmedetomidine and clonidine are viable adjuncts to local anesthetics that offer a faster onset and a better quality of analgesia for patients requiring labor analgesia. However, the relative effectiveness of these adjunctive agents for labor analgesia have not been compared head-to-head. Better data on how these adjuncts compare with each other for labor analgesia efficacy, can result in more informed clinical care strategies.

This trial was initially initiated as a superiority design. After further scientific input, it was decided that a non-inferiority design would be more informative for the clinical question at hand. The hypothesis is that clonidine (Group C) and dexmedetomidine (Group D) are non-inferior to fentanyl (Group F) (usual care) as adjuncts for epidural labor analgesia. The null hypothesis is that clonidine and dexmedetomidine are inferior to fentanyl as adjuncts for epidural labor analgesia. Clinical Protocol specific methodology did not change throughout the trial and the full trial protocol document can be found in the relevant section below. An updated statistical analysis plan includes updated sample size calculations and has been reported to account for the noninferiority analysis plan. No data was analyzed prior to the completion of all data collection procedures.

ELIGIBILITY:
Pregnant minors were not enrolled in this trial.

Inclusion Criteria:

* Pregnant women greater than 18 years of age
* American Society of Anesthesiologists (ASA) Physical Status 2 or 3
* Term pregnancy (greater than 37 gestational weeks)
* Planning epidural labor analgesia
* Singleton pregnancy
* Vertex presentation
* Planned vaginal delivery

Exclusion Criteria:

* Pre-eclampsia with or without severe features
* New initiation of antihypertensive agent within 24 hours prior to enrollment
* Uncontrolled systemic comorbidities [i.e., diabetes, hepatic, renal or cardiac]
* Known or suspected fetal abnormalities
* Allergy to study agents
* Contra-indication to neuraxial anesthesia
* Inability to communicate or participate in study procedures

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant flow numbers reflect mother-fetus dyads (1 mother + 1 infant per dyad). Intervention groups were assigned at the maternal level.
Pre-assignment Details: Pregnant subjects were enrolled at the time of admission to labor and delivery. Both mothers and infants were considered enrolled for the purpose of capturing specific infant information from the infant medical record after delivery (i.e., Apgar scores, cord gases). However, only mothers received the study medication for labor pain control. All other outcomes were assessed on maternal subjects only. Enrollment number & number of subjects started/completed represents the number of dyads enrolled.
Groups:
- Clonidine: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Clonidine 60 mcg
  Clonidine: Clonidine belongs to the drug classification of antihypertensives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
  Pregnant subjects were enrolled at the time of admission to labor and delivery. Both mothers and infants were considered enrolled for the purpose of capturing specific infant information from the infant medical record after delivery (i.e., Apgar scores, cord gases). However, only mothers received the study medication for labor pain control. All other outcomes were assessed on maternal subjects only. Enrollment number & number of subjects started/completed represents the number of dyads enrolled.
- Dexmedetomidine: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Dexmedetomidine 30 mcg
  Dexmedetomidine: Dexmedetomidine belongs to the drug classification of sedatives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
  Pregnant subjects were enrolled at the time of admission to labor and delivery. Both mothers and infants were considered enrolled for the purpose of capturing specific infant information from the infant medical record after delivery (i.e., Apgar scores, cord gases). However, only mothers received the study medication for labor pain control. All other outcomes were assessed on maternal subjects only. Enrollment number & number of subjects started/completed represents the number of dyads enrolled.
- Ropivacaine + Fentanyl: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Fentanyl 100mcg
  Fentanyl: Fentanyl belongs to the drug classification of analgesic opioid agonists and is used as the standard of care
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
  Pregnant subjects were enrolled at the time of admission to labor and delivery. Both mothers and infants were considered enrolled for the purpose of capturing specific infant information from the infant medical record after delivery (i.e., Apgar scores, cord gases). However, only mothers received the study medication for labor pain control. All other outcomes were assessed on maternal subjects only. Enrollment number & number of subjects started/completed represents the number of dyads enrolled.
Period: Overall Study
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Started | 30 (30 mothers, 30 infants) | 29 (29 mothers, 29 infants) | 29 (29 mothers, 29 infants)
Completed | 24 (24 mothers, 24 infants) | 22 (22 mothers, 22 infants) | 23 (23 mothers, 23 infants)
Not Completed | 6 | 7 | 6

BASELINE CHARACTERISTICS:
Population: Baseline data were derived from maternal subjects at the time of enrollment. Baseline data were not collected from fetuses (because enrollment and the study medication administration occurred during pregnancy).
Groups:
- Clonidine (Maternal): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Clonidine 60 mcg
  Clonidine: Clonidine belongs to the drug classification of antihypertensives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
- Dexmedetomidine (Maternal): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Dexmedetomidine 30 mcg
  Dexmedetomidine: Dexmedetomidine belongs to the drug classification of sedatives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
- Ropivacaine + Fentanyl (Maternal): Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Fentanyl 100mcg
  Fentanyl: Fentanyl belongs to the drug classification of analgesic opioid agonists and is used as the standard of care
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
- Total: Total of all reporting groups
Arm/Group | Clonidine (Maternal) | Dexmedetomidine (Maternal) | Ropivacaine + Fentanyl (Maternal) | Total
Number analyzed (Participants) | 24 | 22 | 23 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 23 | 69
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (4.1) | 32 (3.5) | 31.5 (3.9) | 31.33 (3.83)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only female participants.
  Participants
    Female | 24 | 22 | 23 | 69
    Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Burden, AUC (30 Minutes)
Description: Pain score AREA UNDER THE CURVE (AUC), which is a calculated area under curve using the trapezoidal rule, where pain scores measured from 0 (no pain) to 10 (worst imaginable pain) are on the y axis, and time is on the x axis (pain scores were measured at 5 minutes, 10 minutes,15 minutes, 30 minutes after epidural initiation for the primary outcome assessment). The scale for AUC is not 0-10 but rather is completely dependent upon the area generated under the curve created by pain scores for the first 30 minutes of epidural analgesia (primary outcome time frame): in this case, the scale is 0-250 pain units*minute, given maximum pain score possibility of 10 and time period of 30 minutes. The units of AUC are the units of Y axis times units of X axis, in this case, pain score units * minutes. Pain AUC was compared between Fentanyl, Clonidine and Dexmedetomidine groups.
Time Frame: First 30 minutes of analgesia
Population: Maternal only
Measure: Median (Inter-Quartile Range); unit: pain units*minutes
Groups:
- Clonidine: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Clonidine 60 mcg
  Clonidine: Clonidine belongs to the drug classification of antihypertensives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
- Dexmedetomidine: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Dexmedetomidine 30 mcg
  Dexmedetomidine: Dexmedetomidine belongs to the drug classification of sedatives
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
- Ropivacaine + Fentanyl: Bolus dose at epidural initiation, through the epidural catheter:
  10 ml Ropivacaine 0.1 % combined with a single dose of Fentanyl 100mcg
  Fentanyl: Fentanyl belongs to the drug classification of analgesic opioid agonists and is used as the standard of care
  Ropivacaine: Ropivacaine belongs to the drug classification of local or regional anesthesia for surgery and is used as standard of care
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
pain units*minutes | 101 [38 to 138] | 67 [41 to 100] | 39 [22 to 72]
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Non-Inferiority — The noninferiority margin δ was set as the median of fentanyl group + 30 representing a 1-point pain numeric rating scale difference per unit time across the 30-minute initiation period. A conventional 1-sided 95% confidence interval (CI) was constructed using normal distribution assumptions. Analysis was by intent to treat. Comparisons of PI-AUC30 between the three agents were made by one-way ANOVA; p = 0.226, ANOVA

2. Secondary Outcome: Pain Burden, AUC (120 Minutes)
Description: Pain score AREA UNDER THE CURVE (AUC), which is a calculated area under curve using the trapezoidal rule, where pain scores measured from 0 (no pain) to 10 (worst imaginable pain) are on the y axis, and time is on the x axis (pain scores were measured at 5 minutes, 10 minutes,15 minutes, 30 minutes, 60 minutes, 90 minutes and 120 minutes after epidural initiation). The scale for AUC is not 0-10 but rather is completely dependent upon the area generated under the curve created by pain scores for the first 120 minutes of epidural analgesia: in this case, the scale is 0-850 pain units*minute, given maximum pain score possibility of 10 and time period of 120 minutes. The units of AUC are the units of Y axis times units of X axis, in this case, pain score units * minutes. Pain AUC was compared between Fentanyl, Clonidine and Dexmedetomidine groups.
Time Frame: First 120 minutes of analgesia
Population: Maternal only
Measure: Mean (Inter-Quartile Range); unit: pain units*minutes
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
pain units*minutes | 133 [38 to 217] | 67 [41 to 154] | 45 [28 to 132]
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.16, ANOVA

3. Secondary Outcome: Pain Scores
Description: Pain as defined by the Numeric Rating Score (NRS) in which the minimum score of 0 indicates no pain at all and the maximum score of 10 indicates the worst pain imaginable.
Time Frame: 15 minutes after initiation of epidural analgesia
Population: Maternal only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
score on a scale | 2.8 (2.7) | 1.9 (2.5) | 1.0 (1.5)
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.03, ANOVA

4. Secondary Outcome: Pain Scores
Description: as for outcome 3
Time Frame: 30 minutes after initiation of epidural analgesia
Population: Maternal only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
score on a scale | 2.0 (2.4) | 0.9 (2.0) | 0.8 (1.2)
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.07, ANOVA

5. Secondary Outcome: Pain Scores
Description: as for outcome 3
Time Frame: Immediately after delivery
Population: Maternal only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
score on a scale | 1.7 (2.8) | 0.8 (2.3) | 0.5 (0.9)
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.22, ANOVA

6. Secondary Outcome: Cesarean Delivery
Description: This will be measured by yes/no response to cesarean delivery mode of delivery outcome. We report the raw numbers of patients who did receive a cesarean delivery according to group.
Time Frame: At the time of delivery
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 3 | 1 | 3
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.28, Fisher Exact

7. Secondary Outcome: Hypotension
Description: This is measured as any hypotensive event occurring any time between 0-120 min after study drug administration.
Time Frame: Between 0-120 min after study drug administration
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 13 | 10 | 11
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.83, Fisher Exact

8. Secondary Outcome: Nausea
Description: Patient self-report of nausea at any time between 0-120 min after study drug administration
Time Frame: 0-120 min after study drug administration
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 5 | 4 | 5
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.01, Fisher Exact

9. Secondary Outcome: Vomiting
Description: Patient self-report of vomiting at any time between 0-120 min after study drug administration
Time Frame: 0-120 min after study drug administration
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 1 | 0 | 1
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.36, Fisher Exact

10. Secondary Outcome: Shivering
Description: Patient self-report of shivering at any time between 0-120 min after study drug administration
Time Frame: 0-120 min after study drug administration
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 6 | 4 | 7
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.36, Fisher Exact

11. Secondary Outcome: Pruritus
Description: Patient self-report of pruritus at any time between 0-120 min after study drug administration
Time Frame: 0-120 min after study drug administration
Population: Maternal only
Measure: Count of Participants; unit: Participants
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
Participants | 3 | 0 | 5
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.54, Fisher Exact

12. Secondary Outcome: Patient Treatment Satisfaction
Description: Patient self-report regarding satisfaction with analgesia on a scale of 1-10; 1 = not satisfied, 10 = the most satisfied.
Time Frame: Immediately after delivery
Population: Maternal only
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
score on a scale | 10 [8 to 10] | 10 [9 to 10] | 10 [8 to 10]
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.58, Kruskal-Wallis

13. Secondary Outcome: Newborn Apgar Score
Description: The Apgar score is a method of assessing newborn health at the time of delivery. Score range 0 to 10 where 0 is poor health and 10 is the best health.
Time Frame: 1 minute after delivery
Population: Neonatal only
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clonidine | Dexmedetomidine | Ropivacaine + Fentanyl
Number analyzed (Participants) | 24 | 22 | 23
score on a scale | 9 [8 to 9] | 8 [8 to 9] | 8.5 [8 to 9]
Statistical Analysis 1: Comparison: Clonidine vs Dexmedetomidine vs Ropivacaine + Fentanyl; Test type: Superiority; p = 0.98, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From enrollment until 3 days after delivery.
Description: Definition of adverse event and/or serious adverse event used to collect adverse event information was per definitions available on clinicaltrials.gov.
Groups:
- Clonidine (Fetal-neonatal); Dexmedetomidine (Fetal-neonatal); Ropivacaine + Fentanyl (Fetal-neonatal): Per maternal. Study drug was given during pregnancy while uteroplacental perfusion remained intact. Monitoring for AE/SAE for fetus and infant occurred during labor and delivery (fetal safety monitoring) as well as from day 0 through 3 of life (neonatal safety monitoring).
Arm/Group | Clonidine (Maternal) | Dexmedetomidine (Maternal) | Ropivacaine + Fentanyl (Maternal) | Clonidine (Fetal-neonatal) | Dexmedetomidine (Fetal-neonatal) | Ropivacaine + Fentanyl (Fetal-neonatal)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/30 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/29 | 0/30 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 18/30 | 10/29 | 19/29 | 1/30 | 0/29 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine (Maternal) (N=30) | Dexmedetomidine (Maternal) (N=29) | Ropivacaine + Fentanyl (Maternal) (N=29) | Clonidine (Fetal-neonatal) (N=30) | Dexmedetomidine (Fetal-neonatal) (N=29) | Ropivacaine + Fentanyl (Fetal-neonatal) (N=29)
Prolonged Deceleration (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One dyad had a prolonged deceleration documented around 17h10 (01/26/2023). Fetal heart tones were down to 70-90 from baseline of 120 for 7 min. Condition o called and maternal terbutaline was given to decrease uterine tone. Event resolved completely
Maternal Nausea (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Patient self-report of nausea at any time between 0-120 min after study drug administration
Maternal Vomiting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Patient self-report of vomiting at any time between 0-120 min after study drug administration
Maternal Shivering (Nervous system disorders) | 8 (12) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) — Patient self-report of shivering at any time between 0-120 min after study drug administration
Maternal Pruritus (Nervous system disorders) | 1 (1) | 0 (0) | 16 (28) | 0 (0) | 0 (0) | 0 (0) — Patient self-report of pruritus at any time between 0-120 min after study drug administration
Maternal Hypotension (Nervous system disorders) | 13 (13) | 10 (10) | 11 (11) | 0 (0) | 0 (0) | 0 (0) — This is measured as any hypotensive event occurring any time between 0-120 min after study drug administration.

LIMITATIONS AND CAVEATS:
The primary limitation of this study is related to the clonidine and dexmedetomidine doses used for analgesia initiation. The doses were chosen based on what was available in existing literature and clinical experience. Another limitation is that many patients who were eligible and approached declined participation, citing lack of interest in research or primarily a desire to receive only current institutional standards for epidural labor analgesia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT05487196/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT05487196/SAP_003.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT05487196/ICF_002.pdf